CLINICAL TRIAL: NCT05443919
Title: An Exploratory Study to Evaluate the Safety and Efficacy of a Novel Transcatheter Pulmonary Thrombectomy System Which Named 'TwiFlow' for Acute Pulmonary Embolism
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of TwiFlow-System for Acute Pulmonary Embolism
Acronym: TwiFlow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Morningside (Nantong) Medical Co.,Ltd (Other)
Collaborators: Xiamen Cardiovascular Hospital, Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHENXING-2022-02
Record Dates: First submitted 2022-06-23; First posted 2022-07-05 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): The arm contains patients with acute pulmonary embolism who undergoing interventional therapy with transcatheter pulmonary embolectomy system which named 'TwiFlow-Thrombectomy Catheter System'
  Interventions: Device: TwiFlow-Thrombectomy Catheter System

INTERVENTIONS:
Device: TwiFlow-Thrombectomy Catheter System — Patients with acute pulmonary embolism and meeting the conditions of this clinical trial will accept the pulmonary embolism removal operation by the novel device named 'TwiFlow-Thrombectomy Catheter System'.

SUMMARY:
For a prospective, single-arm clinical study, this study plans to recruit patients with acute pulmonary intravascular embolization, use production of transcatheter pulmonary artery bolt system which named 'TwiFlow-Thrombectomy Catheter System' developed by the MorningSide (NanTong) medical device Co., LTD. on pulmonary artery interventional therapy, for evaluating the efficacy and safety of this novel system in the treatment of patients with pulmonary intravascular embolization disease.

DETAILED DESCRIPTION:
As a prospective, single-arm clinical study, the investigators plan to evaluate the new production's efficacy and safety which named 'TwiFlow-Thrombectomy Catheter System'. This study will be carried out in Xiamen Cardiovascular Hospital, Xiamen University. A total of 3 subjects are planned to be enrolled. After screening, all subjects will be treated with transcatheter pulmonary artery thrombectomy system, and clinical follow-up will be conducted at 48 hours, 14 days and 30 days after surgery.

Right Ventricular/Left Ventricular decline from baseline to 48 hours after surgery and the incidence of major adverse events (MAE) within 48 hours after surgery were used as primary endpoints. In instrument performance evaluation, the success rate of surgery, postoperative immediate target lesion embolus removal efficiency, pulmonary artery pressure changes before and after operation value, values of arterial oxygen partial pressure changes before and after operation, death rates related to the equipment in 48 hours after surgery, incident rate of bleeding in 48 hours after operation, postoperative clinical deterioration rate in 48 hours after surgery, postoperative pulmonary vascular injury incidence in 48 hours after surgery, the incidence of heart damage injury in 48 hours after surgery, all-cause death rate in 30 days after surgery, and symptomatic Pulmonary Embolization recurrence rate in 30 days after surgery were secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. 18≤ age ≤75, no gender limitation;
2. patients clinically diagnosed as acute pulmonary embolism requiring pulmonary artery thrombosis clearance;
3. RV/LV ratio ≥0.9;
4. Patients who agreed to participate in the study and voluntarily signed the informed consent.

Exclusion Criteria:

1. Target vessel diameter < 6.6mm;
2. Calcification, plaque or stenosis of target lesions;
3. Hematocrit < 28%;
4. Patients with a history of chronic pulmonary hypertension;
5. Patients with left bundle branch block;
6. A history of chronic left heart failure and left ventricular ejection fraction ≤30%;
7. Patients with abnormal renal function (serum creatinine > 1.8 mg/dL or >159 umol/L);
8. Patients with known coagulopathy or bleeding tendency (platelet <100×109/L, or INR> 3);
9. Patients who cannot receive antiplatelet or anticoagulant therapy;
10. Patients who underwent cardiovascular or pulmonary open surgery within 7 days before surgery;
11. Patients with intracardiac thrombosis;
12. Patients treated with extracorporeal membrane oxygenation;
13. Patients known to be allergic to contrast agents;
14. Patients with diseases that may cause difficulty in treatment and evaluation (such as malignant tumor, acute infectious disease, sepsis, general condition that cannot tolerate surgery, life expectancy less than one year, etc.);
15. Pregnant and lactating women;
16. Patients who are participating in clinical trials of other drugs or medical devices;
17. Other patients deemed unsuitable for the study by the investigator;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Right Ventricular/Left Ventricular decline from baseline to 48 hours after surgery | before and 48 hours after surgery
  Right Ventricular (RV) and Left Ventricular (LV) were recorded during the screening period and 48 hours after surgery by echocardiography or pulmonary artery CT (CTPA), and RV/LV and RV/LV reduction were calculated. The target RV/LV reduction from baseline to 48 hours after surgery was at least 0.2
The incidence of major adverse events (MAE) within 48 hours after surgery | 48 hours after surgery
  The incidence of major adverse events (MAE) during and 48 hours after surgery was observed and recorded, and the incidence of MAE was calculated (referring to the definition of MAE). The target incidence of MAE 48 hours after surgery was less than 25%.
  MAE events defined as those occurring within 48 hours of treatment include device-related death, massive bleeding, pulmonary vascular injury, and cardiac injury.
  Haemorrhage: Disabling or life-threatening bleeding, or severe haemodynamic injury.
  Pulmonary vascular injury: Defined as perforation or injury of a major pulmonary artery branch requiring surgical open surgical intervention.
  Cardiac injury: Defined as heart injury requiring surgical open surgical intervention.

SECONDARY OUTCOMES:
instrument performance evaluation | intraoperative period
  Whether the plug remover is delivered to the specified location or not, whether the thrombectomy stent was successfully deployed or not, whether the plug is retracted successfully or not, whether the thrombectomy device safely removed from the body or not. Whether the conveying system delivers to the specified location or not, whether the delivery system safely removed from the body or not.
the success rate of surgery | intraoperative period
  Surgical success was defined as successful thrombectomy without MAE.
postoperative immediate target lesion embolus removal efficiency | before the pulmonary intravascular embolization removal procedure began and after the embolization removal operation end immediately
  Thrombus clearance = (postoperative target vascular diameter - preoperative target vascular diameter)/preoperative target vascular diameter x100%. The thrombus clearance rate of target lesions can be divided into three grades: <50%, 50-90% and > 90% respectively, in which the thrombus clearance rate ≥50% is effective.
pulmonary artery pressure changes before and after operation value | before the pulmonary intravascular embolization removal procedure began and after the embolization removal operation end immediately
  Changes in pulmonary artery pressure before and after operation = postoperative pulmonary artery pressure - preoperative pulmonary artery pressure
values of arterial oxygen partial pressure changes before and after operation | before the pulmonary intravascular embolization removal procedure began and after the embolization removal operation end immediately
  Preoperative and postoperative arterial oxygen partial pressure = postoperative arterial oxygen partial pressure - preoperative arterial oxygen partial pressure
death rates related to the equipment in 48 hours after surgery | 48 hours after surgery
  death rates
incident rate of bleeding in 48 hours after operation | 48 hours after surgery
  incident rate of bleeding
postoperative clinical deterioration rate in 48 hours after surgery | 48 hours after surgery
  Clinical deterioration include instrumentation related events such as unplanned endotracheal intubation, mechanical ventilation, arterial hypotension (>1 hour) or shock, cardiopulmonary resuscitation, significant deterioration of oxygenation, and emergency surgical embolectomy
postoperative pulmonary vascular injury incidence in 48 hours after surgery | 48 hours after surgery
  Pulmonary vascular injury: Defined as perforation or injury of a major pulmonary artery branch requiring surgical open surgical intervention.
the incidence of heart damage injury in 48 hours after surgery | 48 hours after surgery
  Cardiac injury: Defined as heart injury requiring surgical open surgical intervention.
all-cause death rate in 30 days after surgery | 30 days after surgery
  all-cause death
symptomatic Pulmonary Embolization recurrence rate in 30 days after surgery | 30 days after surgery
  patients present with pulmonary embolism again

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhuang, Dr., Study Chair — Xiamen Cardiovascular Hospital, Xiamen University
Locations (1):
- Atrial shunt implant system, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moore K, Kunin J, Alnijoumi M, Nagpal P, Bhat AP. Current Endovascular Treatment Options in Acute Pulmonary Embolism. J Clin Imaging Sci. 2021 Jan 25;11:5. doi: 10.25259/JCIS_229_2020. eCollection 2021. PMID 33598362
- [Background] Villalba L, Nguyen T, Feitosa RL Jr, Gunanayagam P, Anning N, Dwight K. Single-session catheter-directed lysis using adjunctive power-pulse spray with AngioJet for the treatment of acute massive and submassive pulmonary embolism. J Vasc Surg. 2019 Dec;70(6):1920-1926. doi: 10.1016/j.jvs.2019.03.038. Epub 2019 May 27. PMID 31147112
- [Background] Al-Hakim R, Bhatt A, Benenati JF. Continuous Aspiration Mechanical Thrombectomy for the Management of Submassive Pulmonary Embolism: A Single-Center Experience. J Vasc Interv Radiol. 2017 Oct;28(10):1348-1352. doi: 10.1016/j.jvir.2017.06.025. PMID 28941516
- [Background] Sista AK, Horowitz JM, Tapson VF, Rosenberg M, Elder MD, Schiro BJ, Dohad S, Amoroso NE, Dexter DJ, Loh CT, Leung DA, Bieneman BK, Perkowski PE, Chuang ML, Benenati JF; EXTRACT-PE Investigators. Indigo Aspiration System for Treatment of Pulmonary Embolism: Results of the EXTRACT-PE Trial. JACC Cardiovasc Interv. 2021 Feb 8;14(3):319-329. doi: 10.1016/j.jcin.2020.09.053. Epub 2021 Jan 13. PMID 33454291
- [Background] Yasin JT, Davis R, Saemi A, Regunath H, Krvavac A, Saboo SS, Bhat AP. Technical efficiency, short-term clinical results and safety of a large-bore aspiration catheter in acute pulmonary embolism - A retrospective case study. Lung India. 2020 Nov-Dec;37(6):485-490. doi: 10.4103/lungindia.lungindia_115_20. PMID 33154209
- [Result] Wible BC, Buckley JR, Cho KH, Bunte MC, Saucier NA, Borsa JJ. Safety and Efficacy of Acute Pulmonary Embolism Treated via Large-Bore Aspiration Mechanical Thrombectomy Using the Inari FlowTriever Device. J Vasc Interv Radiol. 2019 Sep;30(9):1370-1375. doi: 10.1016/j.jvir.2019.05.024. Epub 2019 Jul 30. PMID 31375449
- [Result] Tu T, Toma C, Tapson VF, Adams C, Jaber WA, Silver M, Khandhar S, Amin R, Weinberg M, Engelhardt T, Hunter M, Holmes D, Hoots G, Hamdalla H, Maholic RL, Lilly SM, Ouriel K, Rosenfield K; FLARE Investigators. A Prospective, Single-Arm, Multicenter Trial of Catheter-Directed Mechanical Thrombectomy for Intermediate-Risk Acute Pulmonary Embolism: The FLARE Study. JACC Cardiovasc Interv. 2019 May 13;12(9):859-869. doi: 10.1016/j.jcin.2018.12.022. PMID 31072507